CLINICAL TRIAL: NCT00533390
Title: Anti-retroviral Efficacy, Tolerance and Other Pharmacologic Interactions of the Non Nucleoside Analog Efavirenz in Association With Rifampicin to Treat Tuberculosis and AIDS
Brief Title: Randomized Clinical Trial to Assess the Efficacy and Safety of Concomitant Use of Rifampicin and Efavirenz 600 X 800mg
Acronym: IPEC-EFV
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of financial support and low inclusion rate
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, Valeria Cavalcanti Rolla, MD, PhD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE-0017.1.009.000-03
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Tuberculosis; HIV Infections
Keywords: efavirenz; tuberculosis; AIDS; rifampicin; efficacy; safety; Treatment Naive
MeSH Terms: conditions — Tuberculosis; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EFAVIRENZ 800mg (Experimental): Efavirenz 800 mg (tablet) PO QD during 5 months associated with two nucleoside analogs during tuberculosis therapy with rifampicin
  Interventions: Drug: efavirenz
- EFAVIRENZ 600mg (Active Comparator): Efavirenz 600 mg (tablet) PO QD during 5 months associated with two nucleoside analogs during tuberculosis therapy with rifampicin
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: efavirenz — 600mg X 800mg QID during TB therapy with rifampicin associated with other antituberculosis drugs in patients concomitant treated for tuberculosis and AIDS
  Other Names: Stocrin; Sustiva

SUMMARY:
Rifampicin is a potent inducer of the CYP450 and decrease the plasmatic concentration of NNRTI and Protease Inhibitors. In our study we are going to compare the 600 an 800mg doses of efavirenz concomitant of rifampicin use to treat tuberculosis. The hypothesis is that the 800 mg dose would be more adequate than the 600mg

DETAILED DESCRIPTION:
The study consist in a open label randomized clinical trial comparing efavirenz 600mg QID versus efavirenz 800mg QID in patients with tuberculosis (treated with regimens including rifampicin) and AIDS diagnosis. The total duration of the study is 6 months for each patient. All eligible patient will be treated with a fist line regimen for tuberculosis according to Brazilian guidelines: rifampicin (600mg QID); isoniazid (400mg QID) e pyrazinamide (2g QID) during 6 months for a weight of 45 kg or more and adapted doses for persons with less than 45 kg. For patients with previous history of TB therapy etambutol 1.200mg QID will be added to the regimen.

Both groups will receive nucleoside reverse transcriptase inhibitors (NRTI)and a non nucleoside transcriptase inhibitor (NNRTI) to treat HIV. The ITRN of first choice will be zidovudine and lamivudine association. Patients presenting contra indication for the use of those drugs will receive others NRTI. The NNRTI is efavirenz (800 or 600mg).

Antiretrovirals will be initiated 30 days after stable TB therapy. In case of adverse events during TB therapy that lead to treatment interruption, the study drugs will be delayed until the 30th day after triple therapy for TB. During HIV therapy NRTI can be changed in case of intolerance

ELIGIBILITY:
Inclusion Criteria:

* Adults with tuberculosis diagnosis, HIV positive.
* Agreement to avoid not allowed drugs during the trial, agreement to participate in the study (informed consent)

Exclusion Criteria:

* Active liver disease
* Pregnancy or breast feeding
* CD4 counts >350

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
proportion of patients with viral load < 80 at the end of tuberculosis therapy proportion of adverse events in each group | 6 months

SECONDARY OUTCOMES:
Immunologic reconstitution Genotyping resistance | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Valeria C Rolla, MD DSc, Principal Investigator — Instituto de Pesquisa Clinica Evandro Chagas, Fiocruz; Maria Cristina S Lourenço, MSc, Study Chair — Instituto de Pesquisa Clinica Evandro Chagas, Fiocruz; Flávia M Sant'Anna, MSc, Study Chair — Instituto de Pesquisa Clinica Evandro Chagas, Fiocruz; Mariza G Morgado, DSc, Study Chair — Instituto Oswaldo Cruz, Fiocruz; Pedro E Americano do Brasil, MD MSc, Study Chair — Instituto de Pesquisa Clinica Evandro Chagas, Fiocruz; Carolina S Smaltz, PhD student, Study Chair — Instituto de Pesquisa Clinica Evandro Chagas, Fiocruz; Jose L Teixeira, Pharmacist, Study Chair — Instituto de pesquisa Clinica Evandro Chagas; David J Hadad, PhD, Study Chair — Federal University of Espirito Santo; Reynaldo Dietze, PhD, Study Chair — Federal University of Espirito Santo; Moises Palaci, PhD, Study Chair — Federal University of Espirito Santo
Locations (2):
- Brazil (2):
  - Universidade Federal do Espirito Santo, Vitória, Espírito Santo
  - FIOCRUZ Instituto de Pesquisa Clinica Evandro Chagas, Rio de Janeiro, Rio de Janeiro